CLINICAL TRIAL: NCT05519397
Title: Evaluation of the Role of Immune Checkpoints in Response to Breast Cancer Neoadjuvant
Brief Title: Evaluation of the Role of Immune Checkpoints in Response to Breast Cancer Neoadjuvant Therapy
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD. PhD, Istanbul Training and Research Hospital
Other Study IDs: Breast cancer neoadjuvant
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: immune checkpoints; Locally Advanced; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No response: The breast cancer patients with no response to neoadjuvant therapy
  Interventions: Diagnostic Test: Immune checkpoint measurement
- Moderate response: The breast cancer patients with moderate response to neoadjuvant therapy
  Interventions: Diagnostic Test: Immune checkpoint measurement
- Good response: The breast cancer patients with good response to neoadjuvant therapy
  Interventions: Diagnostic Test: Immune checkpoint measurement

INTERVENTIONS:
Diagnostic Test: Immune checkpoint measurement — Measurement of sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active TGF-β1, CTLA-4, PD-L1, PD-1, Tim-3, LAG-3, Galectin-9

SUMMARY:
Breast cancer is the most common type of cancer in women and the second most common cause of death after lung cancer. In epidemiological studies, its prevalence is 22-26%, and the mortality risk due to breast cancer is around 18%.

It is known that the immune system has an important role in tumor development or tumor destruction. Recent studies have shown that tumor cells acquire escape mechanisms to escape host immunity in the tumor microenvironment.

Studies have reported that immune checkpoints are elevated in many types of cancer and have a poor prognosis. Up or down regulation of immune checkpoints is observed to protect breast cancer cells from the anti-tumor responses of the immune system. There are also immune checkpoints found in plasma in soluble form, and the number of studies evaluating soluble immune checkpoints in cancers is very limited in the literature. Measurement of soluble immune control points is easier than those expressed on the surface, and many markers can be evaluated at the same time. There are very few studies in the literature evaluating soluble immune checkpoints in breast cancer.

The aim of this study is to investigate the role of soluble immune checkpoints in predicting the response to neoadjuvant therapy in locally advanced breast cancers.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women and the second most common cause of death after lung cancer. In epidemiological studies, its prevalence is 22-26%, and the mortality risk due to breast cancer is around 18%. While the classification of malignant breast tumors has traditionally been made according to their histological appearance, some subtypes have been defined according to their molecular features. The different behavior of tumors in the luminal group led to the need to divide this group into subtypes as luminal A and B. The luminal group A, which has the highest prevalence among breast cancers; It includes Her2-negative tumors with low proliferative activity, low mitotic rate and histological grade. The prognosis of patients with luminal A tumors is very good and metastases are mostly limited to bones. Luminal-B tumors have a more aggressive course. The most important difference of this group is that tumors have a high proliferation rate. The breakpoint between luminal A and B is generally accepted as less than 14% of tumor cells showing nuclear Ki67 expression immunohistochemically. In addition, approximately 30% of Her2-positive tumors are immunohistochemically in the luminal B phenotype.

It is known that the immune system has an important role in tumor development or tumor destruction. Recent studies have shown that tumor cells acquire escape mechanisms to escape host immunity in the tumor microenvironment.

Immune checkpoints are important molecules that are on the agenda especially after receiving the Nobel Prize in 2018 and in revealing the relationship between cancer and the immune system. Programmed Cell Death Protein-1 (PD-1) and its ligand, PD-L1, are immune checkpoints that act by inhibiting T cell receptor signal transmission and auxiliary stimuli. T cell immunoglobulin and mucin domain 3 (TIM-3) are mostly expressed on interferon-γ producing T cells, Tregs, dendritic cells, B cells, macrophages, natural killer cells (NK) and mast cells.

Studies have reported that immune checkpoints are elevated in many types of cancer and have a poor prognosis. Up or down regulation of immune checkpoints is observed to protect breast cancer cells from the anti-tumor responses of the immune system. Although many studies have been conducted on immune checkpoints in recent years, a limited number of immune checkpoints which are expressed on the cell surface have been evaluated in each study. There are also immune checkpoints found in plasma in soluble form, and the number of studies evaluating soluble immune checkpoints in cancers is very limited in the literature. Measurement of soluble immune control points is easier than those expressed on the surface, and many markers can be evaluated at the same time. There are very few studies in the literature evaluating soluble immune checkpoints in breast cancer.

The aim of this study is to investigate the role of soluble immune checkpoints in predicting the response to neoadjuvant therapy in locally advanced breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced Breast Cancer patients who will receive neoadjuvant therapy

Exclusion Criteria:

* Known immunodeficiency
* Having a primary malignancy other than breast cancer,
* Pregnancy,
* Patients who refused to participate in the study

Ages: 18 Years to 88 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer limited to females
Study Population: Locally advanced Breast Cancer patients who will receive neoadjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Immune checkpoints | 1 day
  Values in pg/ml of sCD25 (IL-2Ra), 4-1BB, CD27, B7.2 (CD86), Free Active TGF-β1, CTLA-4, PD-L1, PD-L2, PD-1, Tim-3, LAG-3, Galectin-9

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc. Prof, Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gu D, Ao X, Yang Y, Chen Z, Xu X. Soluble immune checkpoints in cancer: production, function and biological significance. J Immunother Cancer. 2018 Nov 27;6(1):132. doi: 10.1186/s40425-018-0449-0. PMID 30482248
- [Background] Li Y, Cui X, Yang YJ, Chen QQ, Zhong L, Zhang T, Cai RL, Miao JY, Yu SC, Zhang F. Serum sPD-1 and sPD-L1 as Biomarkers for Evaluating the Efficacy of Neoadjuvant Chemotherapy in Triple-Negative Breast Cancer Patients. Clin Breast Cancer. 2019 Oct;19(5):326-332.e1. doi: 10.1016/j.clbc.2019.03.008. Epub 2019 Apr 11. PMID 31176611
- [Background] Gershtein ES, Korotkova EA, Vorotnikov IK, Sokolov NY, Ermilova VD, Mochalova AS, Kushlinskii NE. Soluble forms of PD-1/PD-L immune checkpoint receptor and ligand in blood serum of breast cancer patients: association with clinical pathologic factors and molecular type of the tumor. Klin Lab Diagn. 2022 Feb 23;67(2):76-80. doi: 10.51620/0869-2084-2022-67-2-76-80. PMID 35192751